CLINICAL TRIAL: NCT03681756
Title: Development of a Lifestyle Intervention for Korean American Women at Risk for Metabolic Syndrome
Brief Title: WALK Study: Women's Active Living for Koreans Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-24293
Record Dates: First submitted 2018-09-19; First posted 2018-09-24 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Physical Activity; Metabolic Syndrome; Lifestyle, Sedentary
MeSH Terms: conditions — Motor Activity; Metabolic Syndrome; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (No Intervention): Participants will receive an in-person session and an activity monitor
- Group 2 (Experimental): Participants will receive an in-person session, an activity monitor, and social support through BAND
  Interventions: Behavioral: WALK

INTERVENTIONS:
Behavioral: WALK — Walking program
  Arms: Group 2

SUMMARY:
The prevalence of metabolic syndrome (MetS) is a health concern among Asians. Growing evidence indicates that Korean Americans had higher MetS prevalence compared to non-Hispanic Whites, but a culturally and linguistically appropriate lifestyle intervention has not been developed for Korean American middle-aged and older women. Thus, the investigators propose to develop a 4-week lifestyle intervention (Women's Active Living for Koreans (WALK) Study) to increase physical activity (PA) and reduce sedentary behavior for Korean American women.

DETAILED DESCRIPTION:
The purpose of this pilot study is to develop a 4-week lifestyle intervention (Women's Active Living for Koreans (WALK) Study) to increase physical activity (PA) and reduce sedentary behavior for Korean American women. The investigators will assess feasibility and acceptability of the WALK Study and potential efficacy of the WALK Study on outcomes including sedentary behavior and PA.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Korean-speaking Korean American women
* Sedentary lifestyle at work and/or during leisure time
* Aged between 40 and 69; 4) intention to be physically active
* KakaoTalk user

Exclusion Criteria

* Medical conditions or physical problems requiring a special care exercise program
* Known bone or join problems that impair the ability to do moderate physical activity
* Participating in a lifestyle modification program or research study
* Planning a trip out of the U.S. during the next 2 months
* Pregnancy.

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Physical activity | Last 7 days
  Time spent in moderate and vigorous activity

SECONDARY OUTCOMES:
Sedentary behavior | Last 7 days
  Time spent in sedentary activity

CONTACTS AND LOCATIONS:
Overall Officials: Ji Won Choi, RN, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No